CLINICAL TRIAL: NCT03186027
Title: Effect of Coenzyme Q10 Plus NADH Supplementation on the Changes in Fatigue Perception, Sleep Disturbances, Autonomic Function and Health-related Quality of Life in CFS/ME - A Randomized, Placebo-controlled, Double-blind Trial.
Brief Title: Coenzyme Q10 Plus NADH Supplementation in Chronic Fatigue Syndrome/Myalgic Encephalomyelitis
Acronym: CONNeCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Vitae Health Innovation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VITAE 2015
Record Dates: First submitted 2017-05-24; First posted 2017-06-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Chronic Fatigue Syndrome
Keywords: chronic fatigue; Sleep problems; Autonomic dysfunction; Health-Related Quality of Life; Coenzyme Q10; NADH
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Parasomnias; Primary Dysautonomias | interventions — coenzyme Q10; NAD; Phosphoserine; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Active Dietary Supplement: ReConnect (CoQ10 plus NADH) and excipients. ReConnect supplementation (CoQ10: 200mg/day plus NADH 20 mg/day) divided into 2 daily dose (2 tablets/ before breakfast and 2 tablets/ before lunch).
  Excipient Dietary Supplement: Placebo (serine plus vitamin C) Placebo supplementation divided into two daily dose (2 tablets/before breakfast and 2 tablets/ before lunch)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator, care provider and participants do not know which individuals have been assigned in each arm or comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active supplement (CoQ10 plus NADH) (Active Comparator): CFS/ME patients will be randomized to evaluate the effect of oral ReConnect supplementation (CoQ10: 200 mg/day plus NADH: 20 mg/day) taking 4 tablets/day during 8-weeks in term.
  Active supplement based on Coenzyme Q10 plus NADH
  Interventions: Dietary Supplement: Coenzyme Q10 plus NADH
- Phosphoserine plus vitamin C (Placebo Comparator): CFS/ME patients will be randomized to assess the effect of placebo (phospho-serine plus vitamin C) taking 4 tablets/day for 8-weeks in term.
  Placebo: phosphoserine plus vitamin C
  Interventions: Dietary Supplement: phosphoserine plus vitamin C

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 plus NADH — Active arm: Coenzyme Q10 plus NADH CFS/ME patients who will be randomized to measure the effect of oral ReConnect supplementation (CoQ10: 200 mg/day plus NADH 20 mg/day; 4 tablets/day) on changes in the fatigue, sleep problems, autonomic function and HRQoL during 8-weeks in term.
  Intervention: Reconnect
  Arms: Active supplement (CoQ10 plus NADH)
Dietary Supplement: phosphoserine plus vitamin C — Placebo arm: phosphoserine plus vitamin C CFS/ME patients who will be randomized to measure the effect of oral Placebo supplementation (phosphoserine and vit C, 4 tablets/day) on changes in the fatigue, sleep problems, autonomic function and HRQoL during 8-weeks in term.
  Intervention: placebo
  Arms: Phosphoserine plus vitamin C

SUMMARY:
The main aim of the study is to examine the effect of oral CoQ10 plus NADH (Reconnect®) supplementation twice daily for 8-weeks on the changes in fatigue perception, sleep disturbances, autonomic dysfunction and HRQoL assessed by patient-reported outcome measures in CFS/ME.

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome, as known as Myalgic Encephalomyelitis (CFS/ME) is a complex and extremely debilitating chronic condition, with no known cause, no established diagnostic tests, and no universal effective therapy. Its symptoms are mainly unexplained disabling fatigue that lasts for six months or more and that does not improve with rest, worsing with physical and mental activity. It is associated with other concomitant symptoms including muscle pain, post-exertional malaise lasting more than 24h, unrefreshing sleep, autonomic dysfunction and cognitive problems worsing quality of life of sufferers. Previous studies have shown that CFS/ME subjects have a significant decrease in CoQ10 and NADH levels in plasma and peripheral blood mononuclear cells (PBMCs), correlating with symptoms of the condition. Hypothesis: CoQ10 plus NADH administration could be beneficial in the improvement of outcome measures and molecular parameters in CFS/ME individuals.

A total of 282 potentially eligible Caucasian CFS/ME subjects who meet both the 1994 Centers for Disease Control and Prevention/Fukuda's definition and 2003 Canadian case criteria for CFS/ME will be initially enrolled in the study. Those patients who don't meet the inclusion criteria will excluded of the study. All participants will be treatment with ReConnect® containing CoQ10 (50 mg) plus NADH (5 mg) vs. placebo twice daily for 8-weeks in term. Scores for fatigue perception, sleep problems, autonomic dysfunction and QoL will be assess by validated questionnaires of Fatigue Impact Scale (FIS-40), Pittsburgh Sleep Quality Index (PSQI), COMPASS-31 and HRV recording device, and HRQoL (36 item Short Form Health survey), respectively.

The primary outcome is to evaluate the efficacy of oral CoQ10 plus NADH (Reconnect®) supplementation twice daily for 8-weeks on the changes in fatigue perception, sleep problems, autonomic dysfunction and health-related quality of life assessed by outcome measures in CFS/ME subjects.

The secondary outcomes are to examine the effect of oral Reconnect® administration on fatigue perception (assessed by FIS-40), sleep disruption (PSQI), autonomic function (COMPASS-31), Heart Rate Variability (HRV) for measuring R-R intervals by mobile device coupled to the Polar H7 thoracic belt and HRQoL (36-items Short Form Health survey).

ELIGIBILITY:
Inclusion Criteria:

1. Patients female between 18 and 65 years old.
2. Body Mass Index (BMI) ≤ 30 mg/m²
3. Subjects who met the 1994 Centers for Disease Control and Prevention/Fukuda definition and 2003 Canadian diagnostic criteria for CFS/ME.
4. Patients must be able to participate, understand and complete questionnaires in Spanish language.
5. Patients who give a signed informed consent before initiating the study.

Exclusion Criteria:

1. Patients who do not fulfilled the 1994 Centers for Disease Control and Prevention/Fukuda definition and 2003 Canadian criteria for CFS/ME.
2. Patients who are participating in another clinical trial of the same or different nature in the last 30 days prior to inclusion.
3. Any participants who, in the opinion of the principal investigator, may not be able to follow instructions or make a good treatment compliance.
4. Subjects that don't give signed informed consent to participate in the study.
5. Participants who are receiving any drug or banned substances and is expected that withdrawal of some medications/products not allowed in the study involves a significant problem.
6. Participants who are pregnant and/or breastfeeding,
7. Participants with autoimmune disorder, cancer, endocrine and metabolic disorders, rheumatic conditions, multiple sclerosis, psychosis, major depression, cardiovascular disease, hematological conditions, use of oral anticoagulants, smokers or had a history of substance abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 282 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Effect of oral Reconnect ® (CoQ10 plus NADH) supplementation on the changes in core symptoms during 8-weeks in CFS/ME subjects. | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Evaluate the effect of oral Reconnect ® supplementation on the changes in fatigue perception measured by the Fatigue Index Scale-40 (40 items) in all study participants. Items Rate: 0 (no fatigue) to 4 (severe fatigue).

SECONDARY OUTCOMES:
Demographic data and clinical parameters | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Sex
Age of onset of symptoms | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Age at onset of fatigue
Concomitant conditions | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Comorbid illnesses associated with ME/CFS
Height will be measured and reported | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Height in meters
Weight will be measured and reported | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Weight in kilograms
Body Mass Index (BMI) | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Height and Weight will be combined to report BMI in kg/m^2
Sleep Quality | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Pittsburgh Quality of Sleep Index (18 items) for non-refreshing sleep
Autonomic Function | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  COMPASS-31 Questionnaire (31-items) to assess autonomic dysfunction
Heart Rate Variability (HRV) recording device | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Time domain - NN (normal-to-normal R-R interval), HRV index (total number of all NN/ the height of the histogram of all NN), SDNN (standard deviation of the NN), RMSSD (the root mean square of differences of successive NN), NN50 (number of pairs of adjacent NN intervals differing by more than 50 ms in the entire recording) and pNN50(NN50/total number of all NN). Frequency domain - TP (the variance of NN intervals over the temporal segment), VLF(power in very low frequency range; < 0.04 Hz), LF (Power in low frequency range; 0.04~0.15 Hz), HF(Power in high frequency range; 0.15~0.4 Hz).
Health-Related Quality of Life SF36 survey | At the beginning (session 2, week 1), intermedium stage (session 3, week 4) and at the close-up of study (session 4, week 8)
  Short Form-36 Health Survey (36-items) to measure quality of life of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alegre, MD; PhD, Principal Investigator — Vall d'Hebron University Hospital (CFS/ME Clinical Unit)
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alegre J, Roses JM, Javierre C, Ruiz-Baques A, Segundo MJ, de Sevilla TF. [Nicotinamide adenine dinucleotide (NADH) in patients with chronic fatigue syndrome]. Rev Clin Esp. 2010 Jun;210(6):284-8. doi: 10.1016/j.rce.2009.09.015. Epub 2010 May 5. Spanish. PMID 20447621
- [Result] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668
- [Result] Castro-Marrero J, Saez-Francas N, Segundo MJ, Calvo N, Faro M, Aliste L, Fernandez de Sevilla T, Alegre J. Effect of coenzyme Q10 plus nicotinamide adenine dinucleotide supplementation on maximum heart rate after exercise testing in chronic fatigue syndrome - A randomized, controlled, double-blind trial. Clin Nutr. 2016 Aug;35(4):826-34. doi: 10.1016/j.clnu.2015.07.010. Epub 2015 Jul 17. PMID 26212172
- [Result] Castro-Marrero J, Saez-Francas N, Santillo D, Alegre J. Treatment and management of chronic fatigue syndrome/myalgic encephalomyelitis: all roads lead to Rome. Br J Pharmacol. 2017 Mar;174(5):345-369. doi: 10.1111/bph.13702. Epub 2017 Feb 1. PMID 28052319
- [Result] Curriu M, Carrillo J, Massanella M, Rigau J, Alegre J, Puig J, Garcia-Quintana AM, Castro-Marrero J, Negredo E, Clotet B, Cabrera C, Blanco J. Screening NK-, B- and T-cell phenotype and function in patients suffering from Chronic Fatigue Syndrome. J Transl Med. 2013 Mar 20;11:68. doi: 10.1186/1479-5876-11-68. PMID 23514202
- [Result] Castro-Marrero J, Cordero MD, Saez-Francas N, Jimenez-Gutierrez C, Aguilar-Montilla FJ, Aliste L, Alegre-Martin J. Could mitochondrial dysfunction be a differentiating marker between chronic fatigue syndrome and fibromyalgia? Antioxid Redox Signal. 2013 Nov 20;19(15):1855-60. doi: 10.1089/ars.2013.5346. Epub 2013 May 29. PMID 23600892
- See also: Vall d'Hebron University Hospital Research Institute (VHIR) — http://www.vhir.org
- See also: Vall d'Hebron University Hospital (HUVH) — http://www.vhebron.net